CLINICAL TRIAL: NCT04737031
Title: Improving Tobacco Treatment Rates for Outpatient Cancer Patients Who Smoke
Acronym: SPP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Frank Leone, Director, Comprehensive Smoking Treatment Program Professor, Critical Care and Pulmonology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 01921; P50CA244690 (NIH); 843062 (Other: Penn Institutional Review Board)
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Smoking; Tobacco Use; Nicotine Dependence
Keywords: Cancer; Smoking; Tobacco Use; Nicotine Dependence; Tobacco Use Treatment Service
MeSH Terms: conditions — Neoplasms; Smoking; Tobacco Use; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): Clinicians and patients will receive no further interventions beyond usual practice.
- Clinician Nudge (Experimental): Clinicians will receive a nudge via Best Practice Alert within the EMR
  Interventions: Other: Clinician Nudge
- Patient Nudge (Experimental): Patients will receive a message sent through myPennMedicine following establishment of their smoking status.
  Interventions: Other: Patient Nudge
- Clinician and Patient Nudge (Experimental): Both strategies described above will be used.
  Interventions: Other: Clinician Nudge; Other: Patient Nudge

INTERVENTIONS:
Other: Clinician Nudge — Investigators will use the Best Practice Alert functionality within the EMR as the conduit to the point of decision-making. Epic currently "fires" a BPA for each new patient presenting to ACC within the Medical Assistant check-in and vital sign workflow, requiring that medical assistants assess tobacco use status within the past 30 days and satisfy the alert with one of three possible answers. Upon opening the Epic Order tab at a patient's next visit after the screening encounter, clinicians will receive the implementation strategy, placed directly over the order interface. The clinician will be required to "acknowledge" or "opt-out" when presented with the order. Opting-out will require clinicians to acknowledge a reason for opt-out using a checklist or free text.
  Arms: Clinician Nudge; Clinician and Patient Nudge
Other: Patient Nudge — Patients will receive a message sent through myPennMedicine following establishment of their smoking status (at the screening encounter). In all cases, the message will include information specific to the upcoming appointment with the oncology clinician.
  Arms: Clinician and Patient Nudge; Patient Nudge

SUMMARY:
The main purpose of this research study is to evaluate the effectiveness of "nudges" to clinicians, to patients, or to both in increasing Tobacco Use Treatment Service (TUTS) referral and engagement; and to explore clinician, patient, inner setting (e.g., clinic), and outer setting (e.g., payment structures) mechanisms related to TUTS referral and engagement. The investigators will employ rapid-cycle approaches to optimize the framing of nudges to clinicians and patients prior to initiating the trial and mixed methods to explore contextual factors and mechanisms.

The investigators will conduct a four-arm pragmatic cluster randomize clinical trial to test the effectiveness of nudges to clinicians, nudges to patients, or nudges to both in increasing TUTS referral and engagement in cancer patients who smoke, vs. usual care (UC). The investigators hypothesize that each of the implementation strategy arms will significantly increase TUTS referral and engagement compared to UC and that the combination of nudges to clinicians and to patients will be the most effective.

DETAILED DESCRIPTION:
Continued tobacco smoking negatively impacts survival among patients with cancer. Routinely delivered evidence-based tobacco use treatment (TUT) would minimize cancer-specific and all-cause mortality, reduce treatment-related toxicity, and improve quality of life. About 50% of cancer patients who smoked prior to their diagnosis continue to smoke after diagnosis and during treatment. The National Comprehensive Cancer Network, American Society of Clinical Oncology, and American Association for Cancer Research, call for implementation of TUT within oncology care. In 2015, TUT received an "A" recommendation from the US Preventive Services Task Force, given the high level of certainty of resulting benefit. The approval specifically focused on clinicians asking all adults about smoking, prescribing FDA-approved cessation medications for smokers, and offering appropriate behavioral interventions.

Despite the importance of TUT, only half of cancer centers consistently identify patient tobacco use, and few cancer centers employ systematic mechanisms to refer patients to evidence-based cessation services. Acknowledging this gap, the National Cancer Institute (NCI) launched the Cancer Center Cessation Initiative (C3I) as part of the Moonshot to help centers develop effective ways to identify and engage patients who smoke. Penn ISC3 MPI Dr. Schnoll was a member of the NCI advisory board that developed this initiative, and Penn Medicine's Abramson Cancer Center (ACC) was in the first funded cohort. Because clinician expertise in TUT is a known barrier, the initial strategy used an automatic "default" electronic medical record (EMR) referral to the ACC Tobacco Use Treatment Service (TUTS). Engagement increased, but clinicians turned off the default 60% of the time, implicating additional important barriers to change.

This study aims to produce dramatic change within oncology by refining and testing implementation strategies informed by behavioral economics. The investigators' work has identified specific cognitive biases among clinicians and patients that prevent TUTS referral and engagement, including clinician pessimism regarding the ability to help patients stop using tobacco, misconceptions about patient resistance to treatment, and implicit biases regarding the capacity for patients to volitionally alter the course of illness. These motivators are related to clinician willingness to invest effort in help giving and may prevent acquisition of new knowledge and skills. From the patient perspective, several studies identify unique challenges that individuals with cancer face when engaging in tobacco cessation efforts, including low self-efficacy, low perceived benefits of quitting, and perceived risk of treatment. Thus, this study focuses on addressing these barriers, in a pragmatic and innovative way, to increase TUTS referral and engagement in cancer care.

The investigators' objectives are to evaluate the effectiveness of "nudges" to clinicians, to patients, or to both in increasing in TUTS referral and engagement; and to explore clinician, patient, inner setting (e.g., clinic), and outer setting (e.g., payment structures) mechanisms related to TUTS referral and engagement. The investigators will employ rapid-cycle approaches to optimize the framing of nudges to clinicians and patients prior to initiating the trial and mixed methods to explore contextual factors and mechanisms.

The investigators will conduct this study with at least 100 clinicians and at least 900 smokers across Penn Medicine's ACC (the clinician sample size may increase with additional clinicians joining Penn and the patient sample size may be higher given the pragmatic design and delay between determination of eligibility [i.e., patient smokes] and nudge delivery at a subsequent visit). They expect the study to yield essential insights into the effectiveness of nudges as an implementation strategy to speed the uptake of high value evidence-based TUT within cancer care, and to advance the understanding of the multilevel contextual factors that drive response to these strategies. These results will lay the foundation for how cancer care settings can ensure that patients with cancer who smoke are engaged with evidence-based TUT and may lead to a future R01 focused on scaling-up this approach across other cancer centers involved in the C3I.

ELIGIBILITY:
Inclusion Criteria:

Clinician participants must meet the following criteria for inclusion:

1. Currently in practice at an Implementation Lab site (UPHS)
2. Prescribing authority in Pennsylvania (i.e., physician, nurse practitioner, physician assistant)
3. Cared for at least 1 tobacco-using patient in 30 days prior to recruitment
4. English-speaking (messages will be in English)

Patient participants must be diagnosed with cancer and report current tobacco smoking (as assessed by an by any staff collecting vital signs or initially rooming the patients such as nurses, front desk staff, MAs, nursing assistants or technicians during an Index Visit). Patients are considered in the analyzable dataset after their Index Visit and after they have a clinic visit with a clinician in the study at which point a nudge may have been delivered (see steps below).

The process by which patients become eligible for inclusion involves a 3-step algorithm employed in the EMR:

Step 1 - All patients seeking care within the participating Abramson Cancer Center programs are screened for tobacco use status in order to ascertain relevance to the project (i.e., tobacco exposure). This screening encounter need not be a visit with a clinician who is in the cluster randomization.

Step 2 - This step occurs at the first visit with a clinician within the cluster randomization. Note that this might be the same encounter in which screening occurs, but does not have to be. At this visit, all patients identified as current smokers are assigned a hidden (i.e., system) variable, the value of which is based on the clinician they are scheduled to meet during that visit (i.e., cluster membership).

Step 3 - The logic is engaged at the next (third in series) visit, wherein the system variable is used to guide the intervention based on the clinician's cohort. There must be this visit to permit the delivery of the nudges (or not, if in usual care arm). The primary outcome is clinician referral for tobacco cessation through the EHR at this visit. Thus, patients eligible for this study are only those who are screened (and positive for tobacco use) and have completed the two visits in their randomly assigned cluster (clinician clusters are the unit of randomization) during the study period.

Outcomes are assessed at the patient level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2146 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jenssen BP, Schnoll R, Beidas RS, Bekelman J, Bauer AM, Evers-Casey S, Fisher T, Scott C, Nicoloso J, Gabriel P, Asch DA, Buttenheim AM, Chen J, Melo J, Grant D, Horst M, Oyer R, Shulman LN, Clifton ABW, Lieberman A, Salam T, Rendle KA, Chaiyachati KH, Shelton RC, Fayanju O, Wileyto EP, Ware S, Blumenthal D, Ragusano D, Leone FT. Cluster Randomized Pragmatic Clinical Trial Testing Behavioral Economic Implementation Strategies to Improve Tobacco Treatment for Patients With Cancer Who Smoke. J Clin Oncol. 2023 Oct 1;41(28):4511-4521. doi: 10.1200/JCO.23.00355. Epub 2023 Jul 19. PMID 37467454
- [Derived] Jenssen BP, Schnoll R, Beidas R, Bekelman J, Bauer AM, Scott C, Evers-Casey S, Nicoloso J, Gabriel P, Asch DA, Buttenheim A, Chen J, Melo J, Shulman LN, Clifton ABW, Lieberman A, Salam T, Zentgraf K, Rendle KA, Chaiyachati K, Shelton R, Wileyto EP, Ware S, Leone F. Rationale and protocol for a cluster randomized pragmatic clinical trial testing behavioral economic implementation strategies to improve tobacco treatment rates for cancer patients who smoke. Implement Sci. 2021 Jul 15;16(1):72. doi: 10.1186/s13012-021-01139-7. PMID 34266468

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2,146 patients were enrolled in this trial. They were seen by a total of 246 clinicians across 88 clusters. Outcome measures were collected for patients.
Units Other Than Participants: Clusters
Period: Overall Study
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Started (Engaged patients (Intent-to-treat, ITT)) | 490; 22 Clusters | 506; 24 Clusters | 405; 19 Clusters | 745; 23 Clusters
Completed (This was an ITT analysis. All engaged patients (2,146) were included in the analysis, even if they did not complete treatment.) | 490; 22 Clusters (For the "Assigned to Usual Care" arm, treatment visit=0 due to the nature of the intervention design. There are no nudges to be delivered. In other words, treatment is completed with the engaged visit, and there are no additional treatment visits.) | 475; 24 Clusters | 312; 19 Clusters | 518; 23 Clusters
Not Completed | 0; 0 Clusters | 31; 0 Clusters | 93; 0 Clusters | 227; 0 Clusters
Not completed — Patients who did not have a treatment visit | 0 | 31 | 93 | 227

BASELINE CHARACTERISTICS:
Population: The following baseline characteristics are for patients only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge | Total
Number analyzed (Participants) | 490 | 506 | 405 | 745 | 2146
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.7) | 61.2 (12.6) | 62.8 (11.7) | 60.7 (12.6) | 61.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 274 | 164 | 327 | 1003
  Male | 252 | 232 | 241 | 418 | 1143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 10 | 5 | 26 | 45
  Not Hispanic or Latino | 486 | 496 | 400 | 718 | 2100
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 6 | 8 | 3 | 12 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 0 | 3
  Black or African American | 114 | 151 | 86 | 200 | 551
  White | 333 | 318 | 283 | 488 | 1422
  More than one race | 4 | 2 | 5 | 5 | 16
  Unknown or Not Reported | 31 | 25 | 27 | 40 | 123
Region of Enrollment [Number; unit: participants]
  United States | 490 | 506 | 405 | 745 | 2146
Marital Status [Count of Participants; unit: Participants]
  Single | 248 | 244 | 199 | 432 | 1123
  Other | 242 | 262 | 206 | 313 | 1023
Clinician Type (seen by patients) [Count of Participants; unit: Participants]
  Advanced Practice Provider (APP) | 130 | 136 | 140 | 136 | 542
  Physician | 360 | 370 | 265 | 609 | 1604
Clinician Specialty (seen by patients) [Count of Participants; unit: Participants]
  Gynecologic oncology | 8 | 21 | 11 | 0 | 40
  Hematologic oncology | 388 | 402 | 358 | 604 | 1752
  Radiology oncology | 94 | 83 | 36 | 141 | 354
Days between arm assignment and engagement [Mean (Standard Deviation); unit: days] | 68.16 (69.9) | 73.42 (76.1) | 64.84 (66.4) | 72.00 (71.7) | 70.10 (71.40)

OUTCOME MEASURES:

1. Primary Outcome: Penetration (Rate of Referral to TUTS or Medication Prescription)
Description: Defined as the proportion of patients who received either a treatment referral (via the BPA or elsewhere in the EHR workflow) or a prescription for tobacco treatment medication (i.e., nicotine replacement, varenicline, or bupropion)
  Based on workflow issues and recommendations from the trial's Data and Safety Monitoring Board (DSMB), the primary outcome for this trial was adjusted to contain both referrals to TUTS and medication prescriptions.
Time Frame: through study completion, up to one year
Population: Outcome measures were not collected for clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 490 | 506 | 405 | 745
Participants | 66 | 180 | 40 | 222

2. Secondary Outcome: Treatment Engagement Rates (Medication)
Description: Defined as the number of patients who make a pharmacologically-assisted quit attempt using any of the seven pharmacotherapies within 30 days of the initial oncology visit, divided by the total number of referred patients
Time Frame: Up to 30 days following baseline
Population: This outcome was only assessed for patients who were referred to TUTS. Outcome measures were not collected for clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 66 | 180 | 40 | 222
Participants | 52 | 66 | 28 | 88

3. Secondary Outcome: Treatment Engagement Rate (Behavioral)
Description: Defined as the number of patients who receive a quit-line referral or in-person or telephone cessation counseling, divided by the total number of TUTS-engaged patients
Time Frame: Up to 90 days after Repeat Visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 66 | 180 | 40 | 222
Participants | 0 | 131 | 0 | 133

4. Secondary Outcome: Quit Attempt Rate
Description: Defined as the number of TUTS-referred patients who make any quit attempt, divided by the total number of TUTS-referred patients
Time Frame: Up to 90 days after Repeat Visit
Population: This outcome was assessed for patients with whom TUTS staff were able to successfully follow up. Outcome measures were not collected for clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 0 | 18 | 0 | 24
Participants | 0 | 14 | 0 | 18

5. Secondary Outcome: Abstinence Rate
Description: Defined as the total number of TUTS-referred patients self-reporting 7-day point prevalence abstinence at a 90-day follow-up assessment, divided by the total number of TUTS-referred patients
Time Frame: Up to 90 days after Repeat Visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 0 | 18 | 0 | 24
Participants | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: through study completion, up to one year
Description: Adverse events were only monitored for patients, not for clinicians.
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
All-Cause Mortality (participants affected / at risk) | 0/490 | 1/506 | 5/405 | 18/745
Serious Adverse Events (participants affected / at risk) | 0/490 | 0/506 | 0/405 | 0/745
Other Adverse Events (participants affected / at risk) | 0/490 | 0/506 | 0/405 | 0/745

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04737031/Prot_SAP_000.pdf